CLINICAL TRIAL: NCT03234153
Title: Neoadjuvant Immunotherapy With Durvalumab in Combination With Tremelimumab in Patients With Muscle-invasive Bladder Cancer Ineligible for Cisplatin-based Chemotherapy.
Brief Title: Neoadjuvant Immunotherapy With Durvalumab and Tremelimumab for Bladder Cancer Patients Ineligible for Cisplatin
Acronym: NITIMIB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NITIMIB-Trial
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Muscle-invasive Bladder Cancer
Keywords: Muscle-invasive Bladder Cancer; Ineligible for Cisplatin-based Chemotherapy; Durvalumab; Tremelimumab
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Single Arm open-Label prospective Phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Tremelimumab (Experimental): Durvalumab 1500 mg i.v. every 4 weeks in combination with Tremelimumab 75 mg i.v. every 4 weeks for a total of 4 cycles before surgery.
  Interventions: Drug: Durvalumab (Imfinzi); Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab (Imfinzi) — Durvalumab 1500 mg i.v. every 4 weeks in combination with Tremelimumab 75 mg i.v. every 4 weeks for a total of 4 cycles before surgery.
  Other Names: Neoadjuvant Immunotherapy
Drug: Tremelimumab — Tremelimumab 75 mg i.v. in combination with Durvalumab 1500 mg i.v. every 4 weeks every 4 weeks for a total of 4 cycles before surgery.
  Other Names: Neoadjuvant Immunotherapy

SUMMARY:
The trial assess the safety and antitumor activity of the anti-PD-L1 antibody Durvalumab in combination with the anti-CTLA4 antibody Tremelimumab.

DETAILED DESCRIPTION:
Background and Rationale:

The outcome for patients with muscle-invasive bladder cancer treated with surgery alone remains dismal with a 5 year survival rate between 25% to 80% depending on the tumor stage and lymph node status. Cisplatin-based chemotherapy regimens (Methotrexate, Vinblastine, Doxorubicin, Cisplatin ; Cisplatin, Methotrexate, Vinblastine; Gemcitabine/Cisplatin) have demonstrated a modest but absolute benefit in overall survival of 5-8% when administered in the neoadjuvant setting. Therefore, neoadjuvant Cisplatin-based regimens are regarded as a standard of care in treating patients with muscle-invasive bladder cancer. However, bladder cancer is a disease of the elderly and due to age-associated factors (e.g. hearing impaired ≥ grade 2), peripheral neuropathy (≥ grade 2), disease associated impairment of renal function (Glomerular filtration rate < 60 mL/min) and performance status (ECOG ≥ 2) 30 to 50% are ineligible for cisplatin-based chemotherapy regimens. Several combinations with Carboplatin have been tested in single arm, phase II trials in patients ineligible for Cisplatin but no standard regimen has been established for this patient population thus far. The Guidelines of the European association of Urology (EAU) do not recommend any neoadjuvant treatment for Cisplatin-ineligible patients.

The advent of immune checkpoint inhibitors like Durvalumab or Azetolizumab, both antibodies blocking the PD1/PD-L1 interaction, have shown promising results as single agents in terms of response (15-46%) and tolerability in the metastatic setting of bladder cancer.

A trial evaluating the safety, tolerability and antitumor activity of the combination of the immune-checkpoint inhibitors Durvarlumab and the anti-CTLA4 antibody Tremelimumab in various solid tumors, including urothelial carcinoma of the bladder is ongoing (protocol D4190C0010). Blocking the PD1/PD-L1 pathway in combination with an anti-CTLA4 antibody has shown greater antitumor activity than each antibody alone in malignant melanoma trials and showed a promising antitumor activity (17% overall response rate, irrespective of the PD-L1 expression status on tumor cells) in a phase Ib study of metastatic non-small-cell lung cancer. The safety profile was acceptable (42% grade 3-4 treatment related adverse events across all dosing cohorts, most common were diarrhea, colitis and increase lipase), however, the rate of adverse events (e.g. autoimmune phenomena) and treatment interruptions was higher as compared to single agent use.

Objective:

The Primary objective of the trial is to assess the safety and antitumor activity of the anti-PD-L1 antibody Durvalumab in combination with the anti-CTLA4 antibody Tremelimumab.

Study Duration:

Trial study duration encompassed the time from when the participant signs the informed consent until the last protocol-specific procedure has been completed (Cystectomy between week 17 to 23). All patients will be followed up for up to 78 weeks after end of treatment.

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent Form
* ECOG performance status of 0 or 1
* Histologically confirmed muscle-invasive urothelial carcinoma of the bladder (T2-T4 and/or N+). Patients with mixed histologies are required to have a dominant transitional cell pattern.
* Measurable disease according to RECIST v1.1 criteria
* Representative fresh tumor specimen; TURB (transurethral resection of bladder ) specimens must contain a muscle invasive component (at least T2)
* Ineligible to receive cisplatin-based neoadjuvant chemotherapy based on at least one of the following criteria:

  * Creatinin clearance less than 60ml/min (24h urine)
  * CTCAE Gr ≥ 2 hearing loss
  * CTCAE Gr ≥ 2 neuropathy
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Body weight >30 kg
* Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 14 days prior the first study treatment:
* Absolute neutrophil count (ANC) ≥ 1500 cells/µl
* WBC counts > 2500/µl
* Platelet count ≥ 100,000/µl
* Hemoglobin ≥ 9.0 g/dL
* AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 x ULN
* INR and aPTT ≤ 1.5 x ULN
* Serum creatinine clearance (CrCl) ≥ 40 mL/min using the Cockcroft-Gault equation
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for premenopausal female. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

Exclusion Criteria:

* Known metastatic disease
* Intravesical chemo- or biological/immune (BCG) therapy within 6 weeks of first treatment dose
* Prio treatment with immune checkpoint blockade therapies like anti-CTLA-4, anti-PD1 and anti-PD-L1 therapeutic antibodies, including durvalumab and tremelimumab
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis or glomerulonephritis Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this study
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of investigational drug.
* Female patients who are pregnant or breast feeding as well as male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy.
* Known allergy or hypersensitivity to any of the investigational study drugs or any of the study excipients.
* Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Uncontrolled intercurrent illness, including but limited to, ongoing infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina.
* Patients with prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan
* Positive test for HIV
* Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen test at screening) or hepatitis C.
* Active tuberculosis
* Administration of a living, attenuated vaccine within 4 weeks prior to treatment start
* Severe infection within 4 weeks prior to cycle 1, day 1
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior treatment start or anticipated requirement for systemic immunosuppressive medications during the trial. The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids, and mineralocorticoids is allowed
* Known allergy or hypersensitivity to any of the study drugs or any of the study excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 16 weeks
  Response rate (computer tomography or magnet resonance imaging) as measured per standard RECIST v1.1 after four cycles of combined treatment with Durvalumab (MEDI4736) and tremelimumab.

SECONDARY OUTCOMES:
Adverse Events | 26 weeks
  Number of Patients experiencing Toxicity/Adverse Events (AE)
Recurrence-free Survival | 78 weeks
  Number of Patients with Recurrence-free Survival at 78 weeks
Overall Survival | 78 weeks
  Number of Patients alive at 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julian Schardt, MD, Study Chair — Departement of Medical Oncology, University Hospital Berne
Locations (1):
- Departement of Medical Oncology, University Hospital Berne, Bern, Switzerland